CLINICAL TRIAL: NCT07140926
Title: Digital Innovation in Medication-Assisted Treatment for Opioid Use Disorder: A Stepped-Wedge Cluster Randomized Trial
Brief Title: A Stepped-Wedge Cluster Randomized Trial of a Digital App to Support Medication-Assisted Treatment in Individuals With Opioid Use Disorder
Acronym: SMART-OUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bright Therapeutics (Industry)
Collaborators: Community Medical Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 11629
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder
Keywords: Digital Intervention; Opioid Use Disorder; Treatment Retention; Stepped-Wedge Cluster Randomized Trial; Digital Application; Medication-Assisted Treatment; Addictions
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge cluster randomized trial. Clusters of clinics will transition in a randomized sequence from a control period (usual care) to an intervention period (Recovery Connect). Each cluster serves as its own control, allowing comparisons within and across clinics. The stepped-wedge design was chosen to enable pragmatic, real-world implementation while maintaining the ability to assess causal effects. The staggered rollout also allows adjustment for temporal trends and clinic-level variability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Implementation of digital app at the clinic (Recovery Connect) (Experimental): Implementation consists of two components:
  Clinician training: Addiction treatment professionals complete live virtual training with step-by-step guides, video tutorials, and ongoing technical support. Training covers app features, patient linkage, and app-based communication strategies.
  Patient onboarding: Following training, clinicians introduce the app to newly admitted patients, assist with downloading and linking via QR code, and demonstrate core features such as daily check-ins, homework activities, and secure messaging.
  Interventions: Device: Recovery Connect
- Usual Care (No Intervention): Clinics in the control condition continue providing standard medication-assisted treatment (MAT) for opioid use disorder (OUD) without the Recovery Connect app. Usual care includes in-person counseling sessions, medication management, and access to peer support and ancillary services, following each clinic's existing protocols and best practices. Patients do not receive access to the Recovery Connect platform during this phase, and clinicians do not use app-based tools or data to inform care.

INTERVENTIONS:
Device: Recovery Connect — Recovery Connect is a white-labeled version of the Recovery Path platform, rebranded to maintain partner organizations' brand identity while leveraging its established digital infrastructure. Recovery Path is a HIPAA-compliant remote patient monitoring system that supports a blended model of care for medication for opioid use disorder (MOUD), integrating in-person treatment with continuous digital engagement.
  The app provides patients with daily check-ins, access to evidence-based resources and coping strategies, and secure messaging with their care teams. Clinicians receive real-time data on patient progress, risks, and setbacks. Between visits, clinicians can recommend tailored coping tools and psychoeducational content, reinforcing accountability and enhancing continuity of care.
  RC is also integrated into the clinic's electronic medical record system to streamline workflows, reduce administrative burden, and improve documentation accuracy through auto-generated case notes.
  Arms: Implementation of digital app at the clinic (Recovery Connect)

SUMMARY:
The goal of this clinical trial is to learn if a mobile health app called Recovery Connect can help people stay in treatment for opioid use disorder. The study is being done with adults receiving medication-assisted treatment in outpatient opioid treatment programs.

The main questions it aims to answer are:

Does Recovery Connect increase the number of people who remain in treatment after 30 days?

Does Recovery Connect improve continuity of care during the first month of treatment?

Researchers are using a stepped-wedge design, which means that all participating clinics will eventually use the app, but they will begin at different time points in a randomized order. This allows researchers to compare outcomes before and after each clinic starts using Recovery Connect.

Participants will:

Use the Recovery Connect app for daily check-ins, coping strategies, and reminders to support their recovery

Share progress and risk information through the app so counselors can provide timely, personalized support

Work with treatment teams trained to use the app to guide care and reinforce accountability

DETAILED DESCRIPTION:
This study is a stepped-wedge cluster randomized clinical trial evaluating the implementation and effectiveness of Recovery Connect, a mobile health application designed to support individuals receiving medication-assisted treatment (MAT) for opioid use disorder (OUD). Recovery Connect is intended to enhance treatment delivery by:

Providing clinicians with real-time, self-monitored patient progress data to support measurement-based and data-informed care.

Delivering personalized care plans, reminders, and evidence-based coping strategies directly to patients.

Facilitating continuous communication and accountability between patients and counselors between sessions.

Study Design

The trial is conducted across nine outpatient opioid treatment program (OTP) clinics, grouped into eight clusters. Using a stepped-wedge design, each cluster will transition from usual care to the Recovery Connect intervention at randomized, sequential time points, such that all clinics will eventually receive the intervention. All clinicians at each cluster will receive standardized training on Recovery Connect at rollout, with follow-up reinforcement training provided two weeks later. Auxiliary staff (e.g., front desk, peer support, navigators) will also be trained to support patient onboarding.

Participants All clinicians at participating clinics will be included. Patient-level data will be analyzed for all new admissions and readmissions during the study period.

Data Collection

App Usage and Engagement: Patient and clinician usage data, including daily check-ins, logins, and secure messages, will be captured directly through the app.

Patient Treatment Outcomes: Treatment retention and continuity data will be obtained via the Methasoft medical record system, following standard clinic protocols.

Operational Definitions

Exposure: Patients are considered "exposed" if their admission occurred after clinicians at their clinic had completed Recovery Connect training.

Linkage: Patients are considered "linked" if they downloaded the app and were connected with a trained clinician during admission.

Engagement: Defined by app activity within the first week after linkage, including logins, daily check-ins, and secure messaging.

Analyses The primary analyses will use an intent-to-treat framework, including all eligible patients whose clinic underwent Recovery Connect training. Outcomes will be assessed using multilevel logistic regression and cluster-controlled discrete-time survival analyses, accounting for the stepped-wedge design.

ELIGIBILITY:
Inclusion Criteria:

* All newly admitted patients to participating clinics

Exclusion Criteria:

* Dosing suggesting a transfer from a non-participating clinic, or if they had previously used the app prior to their most recent admission during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1524 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment retention | From admission to 60 days post admission (in order to determine whether a 30 day gap began in the first 30 days and thus determine 30-day retention)
  Retention is defined according to federal guidelines, which allow patients to be readmitted within 30 days without restarting the intake process. A patient is considered not retained if a treatment gap of 30 consecutive days begins within the first 30 days after intake. The first day of that gap is recorded as the dropout date.

SECONDARY OUTCOMES:
Treatment continuance | From admission to 30 days post-admission
  Defined as have received at least three quarters (75%) of expected daily doses within the first 30 days following admission, and at least one dose administered during the final week of that period.
3, 7, and 30 day doses | 3, 7 and 30 days post admission
  Number of daily medications for opioid use disorder administered successfully and confirmed, during the first 3, 7 and 30 days post admission.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Palacios, MD, PhD, Principal Investigator — Bright Therapeutics
Locations (9):
- United States (9):
  - Community Medical Services, Anchorage, Alaska
  - Community Medical Services, Wasilla, Alaska
  - Community Medical Services, Billings, Montana
  - Community Medical Services, Bozeman, Montana
  - Community Medical Services, Kalispell, Montana
  - Community Medical Services, Missoula, Montana
  - Community Medical Services, Fargo, North Dakota
  - Community Medical Services, Grand Forks, North Dakota
  - Community Medical Services, Minot, North Dakota

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during this study will not be publicly available due to data confidentiality agreements in place between Bright Therapeutics and Community Medical Services, but select de-identified data will be made available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Palacios JE, Sherrick R, Janssen T, Deuble E, Lorenzen S, Schaefer M, Tregarthen J. Implementation of a Mobile Digital Tool Supporting Medication for Opioid Use Disorder Treatment Improves Retention: Stepped-Wedge Cluster Randomized Controlled Trial. J Med Internet Res. 2025 Dec 22;27:e83346. doi: 10.2196/83346. PMID 41429011